CLINICAL TRIAL: NCT00006002
Title: A Phase II Trial of SU5416 (NSC# 686819) in Patients With Hormone Refractory Prostate Cancer
Brief Title: SU5416 Compared to Dexamethasone in Treating Patients With Progressive Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10428; UCCRC-10428; UCCRC-NCI-49; NCI-49
Record Dates: First submitted 2000-07-05; First posted 2003-08-29 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; Semaxinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm B (Experimental): dexamethasone followed by SU5416 done twice weekly (Monday and Thursday or Tuesday and Friday) every week for 4 weeks (a total of 8 doses). Four weeks of treatment (8 doses) is considered 1 cycle of treatment if tumor grows.
  Interventions: Drug: dexamethasone; Drug: semaxanib
- Arm A (Experimental): SU5416 done twice weekly (Monday and Thursday or Tuesday and Friday) every week for 4 weeks (a total of 8 doses). Four weeks of treatment (8 doses) is considered 1 cycle of treatment
  Interventions: Drug: semaxanib

INTERVENTIONS:
Drug: dexamethasone
  Arms: Arm B
Drug: semaxanib

SUMMARY:
RATIONALE: SU5416 may stop the growth of prostate cancer by stopping blood flow to the tumor. Dexamethasone may be effective in slowing the growth of prostate cancer cells. It is not yet known whether SU5416 or dexamethasone is more effective in treating progressive prostate cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of SU5416 with that of dexamethasone in treating patients who have progressive prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to progression in patients with hormone refractory prostate cancer treated with dexamethasone with or without SU5416.
* Determine the differences in PSA kinetics and PSA hazard score between these two regimens in this patient population.
* Determine the objective response rate and time to development of new lesions in these patients treated with SU5416.
* Determine the toxicity of SU5416 in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral dexamethasone once a day 6 days a week. Treatment continues until disease progression, at which time patients cross over to arm II.
* Arm II: Patients receive oral dexamethasone as in arm I followed by SU5416 IV over 60 minutes twice weekly for 4 weeks. A smaller dose of dexamethasone is administered the day after SU5416. Treatment continues for a minimum of 2 courses in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: A total of 60 patients (30 per arm) will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer not amenable to curative treatment with surgery or radiotherapy
* Progressive disease defined by 1 of the following criteria:

  * New bone scan lesions
  * New or progressive radiologic lesions
  * Sequential increases in PSA on at least 2 successive measurements no less than 2 weeks apart of at least 50% above nadir on prior therapy provided absolute value at time of enrollment is at least 5 ng/mL
* Progressive disease, as defined above, despite adequate hormonal therapy defined by all of the following:

  * Continued treatment with an LHRH agonist or prior orchiectomy
  * Sequential or concurrent treatment with an antiandrogen (e.g., flutamide, nilutamide, or bicalutamide)
  * Trial of antiandrogen withdrawal at least 4 weeks prior to study
* CNS metastasis allowed if:

  * Previously treated
  * Neurologically stable
  * Oral or intravenous steroids or anticonvulsants not required
  * Brain scan (CT or MRI) within the past 2 weeks shows no active or residual disease

    * Negative brain scan required if neurologic signs or symptoms suggestive of CNS metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No uncompensated coronary artery disease
* No history of myocardial infarction or severe unstable angina within the past 6 months
* No severe peripheral vascular disease associated with diabetes mellitus
* No deep venous or arterial thrombosis within the past 3 months

Pulmonary:

* No pulmonary embolism within the past 3 months

Other:

* Not pregnant
* Fertile patients must use effective contraception
* No significant uncontrolled underlying medical or psychiatric illness
* No serious active infection
* No other prior or concurrent malignancy except nonmelanoma skin cancer unless completed therapy and considered to be at less than 30% risk of relapse
* No history of severe allergic or anaphylactic reactions to paclitaxel or docetaxel

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy
* No other concurrent chemotherapy
* No other concurrent investigational antineoplastic drugs

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-06; Primary Completion 2002-09 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (18):
- United States (18):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Division of Hematology/Oncology, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina